CLINICAL TRIAL: NCT05832411
Title: Effect of Artificial Intelligence Monitoring Blind Spots of EGD on the Inspection Time and Dection Rate of Neoplastic Lesions
Brief Title: Effect of AI Monitoring Blind Spots of EGD on the Inspection Time and Lesion Dection Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EA-23-005
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Upper Gastrointestinal Symptoms
Keywords: Esophagogastroduodenoscopy; Artificial intelligence; Blind spot
MeSH Terms: conditions — Scotoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI group (Experimental): In the AI group, except for the original videos, there is additional information presented to endoscopists:（1）the virtual stomach model monitoring;（2）time;（3）scoring. Endoscopists will complete EGD examination without blind spots.
  Interventions: Device: Endoangle
- Routine group (No Intervention): In the Routine group, only the original videos and there is no additional information, and inspection time will be no less than 7 minutes.

INTERVENTIONS:
Device: Endoangle — there is additional information presented to endoscopists:（1）the virtual stomach model monitoring；（2）time;（3）scoring.
  Arms: AI group

SUMMARY:
The goal of this clinic trial is to learn about the effect of AI monitoring blind spots on the inspection time to EGD. Patients are randomly assigned to undergo an EGD with or without the assistance of AI. In the AI group, except for the original videos, there is additional information presented to endoscopists:(1)the virtual stomach model monitoring;(2)time;(3)scoring. Researchers will compare intervention group to see if it have a shorter inspection time compared with the control group.

DETAILED DESCRIPTION:
The goal of this clinic trial is to evaluate the effect of real-time artificial intelligence for monitoring blind spots on the inspection time of EGD. Patients are randomly assigned to undergo an EGD with or without the assistance of AI. In the AI group, except for the original videos, there is additional information presented to endoscopists:(1)the virtual stomach model monitoring;(2)time;(3)scoring. Researchers will compare intervention group to see if it have a shorter inspection time in the case of non-inferior detection rate of gastric neoplastic lesions.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18 years or older
2. patients able to give informed consent
3. American Society of Anesthesiology risk class 1,2 or 3

Exclusion Criteria:

1. patients with absolute contraindications to EGD examination
2. patients with a history of previous gastrectomy
3. patients with a serious underlying disease
4. pregnant patients
5. researchers believe that the patient is not suitable to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1672 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Dection rate of neoplastic lesions | Through study completion, an average of 1 year
  Proportion of patients with neoplastic lesions among all patients undergoing esophagogastroduodenoscopy.

SECONDARY OUTCOMES:
Inspection time | 20min
  It is the time from intubation to extubation of the patient without biopsy.

IPD SHARING:
Plan to Share IPD: No
Sponsor approval for data sharing should be sought; Data access requests should be made via an application form detailing the specific requirements and the proposed research and publication plan

REFERENCES:
- [Background] Wu L, Zhang J, Zhou W, An P, Shen L, Liu J, Jiang X, Huang X, Mu G, Wan X, Lv X, Gao J, Cui N, Hu S, Chen Y, Hu X, Li J, Chen D, Gong D, He X, Ding Q, Zhu X, Li S, Wei X, Li X, Wang X, Zhou J, Zhang M, Yu HG. Randomised controlled trial of WISENSE, a real-time quality improving system for monitoring blind spots during esophagogastroduodenoscopy. Gut. 2019 Dec;68(12):2161-2169. doi: 10.1136/gutjnl-2018-317366. Epub 2019 Mar 11. PMID 30858305
- [Background] Wu L, Xu M, Jiang X, He X, Zhang H, Ai Y, Tong Q, Lv P, Lu B, Guo M, Huang M, Ye L, Shen L, Yu H. Real-time artificial intelligence for detecting focal lesions and diagnosing neoplasms of the stomach by white-light endoscopy (with videos). Gastrointest Endosc. 2022 Feb;95(2):269-280.e6. doi: 10.1016/j.gie.2021.09.017. Epub 2021 Sep 20. PMID 34547254
- [Background] Bisschops R, Areia M, Coron E, Dobru D, Kaskas B, Kuvaev R, Pech O, Ragunath K, Weusten B, Familiari P, Domagk D, Valori R, Kaminski MF, Spada C, Bretthauer M, Bennett C, Senore C, Dinis-Ribeiro M, Rutter MD. Performance measures for upper gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2016 Sep;48(9):843-64. doi: 10.1055/s-0042-113128. Epub 2016 Aug 22. No abstract available. PMID 27548885
- [Derived] Tan X, Yao L, Dong Z, Li Y, Yu Y, Gao X, Zhu K, Su W, Yin H, Wang W, Luo C, Li J, You H, Hu H, Zhou W, Yu H. Artificial Intelligence as a Surrogate for Inspection Time to Assess Completeness in Esophagogastroduodenoscopy: A Prospective, Randomized, Noninferiority Study. Clin Transl Gastroenterol. 2025 Mar 25;16(6):e00839. doi: 10.14309/ctg.0000000000000839. eCollection 2025 Jun 1. PMID 40125855